CLINICAL TRIAL: NCT07256756
Title: A Phase I Study of Engineered Tumor Infiltrating Lymphocytes Injection (GC203 TIL) in Patients With Advanced Solid Tumors
Brief Title: A Study of GC203 TIL in Advanced Solid Tumors (NF)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Collaborators: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC203-2025-NF-ST
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC203 TIL (Experimental): participants with advanced solid tumors using cryopreserved GC203 TIL
  Interventions: Biological: GC203 TIL

INTERVENTIONS:
Biological: GC203 TIL — A tumor sample is resected from each participant and cultured ex vivo to expand the population of engineered tumor infiltrating lymphocytes injection (GC203 TIL). After lymphodepletion, patients are infused GC203 TIL.

SUMMARY:
This study is a prospective, open-label, single-arm clinical trial aimed at evaluating the safety and efficacy of GC203 TIL therapy in treating malignant solid tumors that have failed standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* have one the tumor resection for gene-edited GC203 TIL production and successfully produced；
* Age: 18 years to 75years;
* Histologically diagnosed as solid tumor;
* Expected life-span more than 3 months;
* ECOG score 0-1;
* Test subjects have failed standard treatment regimens, and be willing to receive engineered GC203 TIL therapy;
* At least 1 evaluable tumor lesion;

Exclusion Criteria:

* with other malignant tumors,except for the malignancies that have been cured, have been inactive for ≥5 years prior to study inclusion and have a very low risk of recurrence; Non-melanoma skin cancer or malignant lentigo with adequate treatment and no evidence of disease recurrence; Carcinoma in situ with adequate treatment and no evidence of disease recurrence;
* Need glucocorticoid treatment, and daily dose of Prednisone greater than 10mg(or equivalent doses of hormones) or outoimmune diseases requiring immunomodulatory treatment;
* Breathe indoor air in a quiet state, and the oxygen saturation of finger pulse is < 95%;
* Human immunodeficiency virus (HIV) infection or anti-HIV antibody positive, active HBV or HCV infection (HBsAg positive and/or anti-HCV positive), syphilis infection or Treponema pallidum antibody positive;
* Significant cardiovascular anomalies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 month
  To characterize the safety profile of GC203 TIL in patients with Solid Tumors who were failed to standard treatment as assessed by incidence of adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  Proportion of patients with response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Disease Control Rate (DCR） | Up to 36 months
  Proportion of patients with response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Duration of Response (DOR) | Up to 36 months
  The time length between the first confirmed objective response per RECIST 1.1 to the treatment and the subsequent disease progression per RECIST 1.1
Progression-Free Survival (PFS) | Up to 36 months
  The time from TIL infusion until disease progression or death from any cause.
Overall Survival(OS) | Up to 36 months
  The time from TIL infusion until death from any cause.